CLINICAL TRIAL: NCT05537389
Title: Central Lines Filtration in Newborns: a Multicenter Randomized Controlled Trial
Brief Title: Intravenous Neonatal Central Access Safety Trial
Acronym: INCAS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Collaborators: Pall Corporation (Other)
Responsible Party: Principal Investigator, Francesco Cresi, MD, PhD, Study Director, University of Turin, Italy
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: INCAS
Record Dates: First submitted 2022-09-09; First posted 2022-09-13 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Newborn Complication; Catheter Complications

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Patients with central venous access (central umbilical venous catheter or epicutaneous cava catheter)
- Filter (Experimental): Patients with central venous access and in-line filters (central umbilical venous catheter or epicutaneous cava catheter)
  Interventions: Device: In-line filter

INTERVENTIONS:
Device: In-line filter — All infusions, with the exception of some solutions (eg blood products), will be subjected to filtration. The aqueous solutions (parenteral therapy and drugs) will be administered through 0.2 μm filters which will be replaced every 96 h; the lipid emulsions will be administered through 1.2 μm filters which will be replaced every 24 h.
  In case of emergency, life-saving drugs will be administered with bolus modality though the infusion line closer to the patient without the need for filtration.
  In case of drugs/solutions not supported by filtration (eg blood products), they will be administered through a dedicated unfiltered access, which will be removed as soon as the drug is no longer needed.
  Arms: Filter

SUMMARY:
Particulate contamination due to infusion therapy (administration of parenteral nutrition and medications) carries a potential health risk for infants in neonatal intensive care units (NICU).

In-line filtration is increasingly used in critically-ill infants but its benefits, by preventing micro-particle infusion in neonates, remain to be demonstrated.

In-line filters in the intravenous administration sets prevent the infusion of particles, which may reduce infectious complications.

DETAILED DESCRIPTION:
BACKGROUND Particulate contamination due to infusion therapy (administration of parenteral nutrition and medications) carries a potential health risk for infants in neonatal intensive care units (NICU).

This particulate consists of metals, drug crystals, glass fragments or cotton fibres and can be generated by drug packaging, incomplete reconstitution and chemical incompatibilities.

Filters have been shown to remove micro-organisms, endotoxin, air and particles in critically-ill adults and older infants, but its benefits in newborn remain to be demonstrated.

Although recommendations for the use of in-line intravenous filters have been published, there is no consensus on their use.

Moreover, 50% of inflammatory episodes in the setting of NICU are blood culture-negative. These episodes could be partly related to the presence of particles in the infusion lines.

PROJECT AIMS AND DESIGN:

Aim of this multicenter trial is to evaluate the effectiveness of in-line filtration in reducing culture-negative inflammatory episodes in infants admitted to NICU. Further aim is to evaluate the efficacy in the reduction of main CVC-associated complications when using filters.

PATIENTS:

All infants admitted to the NICUs are considered eligible for inclusion into the trial if prolonged infusion therapy (one week or more) is expected, with either umbilical vein catheters (UVC) in a central position or percutaneously inserted central venous catheter. Infants in whom a peripheral UVC is placed but for whom infusion therapy via central venous access is planned will be enrolled too.

Exclusion criteria: Infants will be excluded from participation in the trial if they have clinical characteristics requiring transfer to units not participating in the study before discontinuation of infusion therapy (neurological or surgical diseases, chromosomal abnormalities, and major malformations)..

PROTOCOL:

After randomization each infant will be subsequently allocated to experimental group (Filter) or to control group (Control) as per randomization. Each research unit will refer to its own protocols for infection sulveillance and prevention, although respecting some minimal standard criteria and indications, common and approved by all research units.

In the filter group, all infusions, with the exception of some solutions (eg blood products), will be subjected to filtration. The aqueous solutions (parenteral therapy and drugs) will be administered through 0.2 μm filters which will be replaced every 96 h; the lipid emulsions will be administered through 1.2 μm filters which will be replaced every 24 h. In case of emergency, life-saving drugs will be administered with bolus modality though the infusion line closer to the patient without the need for filtration. In case of drugs/solutions not supported by filtration (eg blood products), they will be administered through a dedicated unfiltered access, which will be removed as soon as the drug is no longer needed.

In the control group, all infusion will be administered through unfiltered accesses.

Data will be collected daily from enrolment up to 48 h after discontinuation of infusion therapy.

In case of inflammatory episode, all patients will undergo to defined specimens, as always in correct clinical practice: complete blood count, sepsis biomarkers (C- reactive protein, procalcitonin, presepsin) and blood culture.

At discharge information regarding the main neonatal pathologies will be recorded.

MAIN OUTCOME Frequency of patients with at least one inflammatory episode sepsis-like, defined by alteration of the biomarkers of inflammation in a negative-culture contest.

SECONDARY OUTCOMES

* Frequency of patients with at least one inflammatory episode defined by alteration of the biomarkers of inflammation in a positive-culture contest.
* Occurrence of phlebitis or local cutaneous inflammation
* Occurrence of luminal obstruction and/or extravascular fluid effusion
* Duration of mechanical ventilation
* Number of catheter days
* Length of stay
* Neonatal mortality

SAMPLE SIZE:

The baseline risk of inflammatory states in the target population remains undetermined. However, we hypothesize a range between 30% and 35%. Consequently, a median risk of 32.5% was assumed for the control group. With the application of filters, a plausible 30% risk reduction is anticipated, resulting in an estimated risk of 22.75% in the intervention arm. Utilizing Fisher's exact test to compare two independent proportions, with an alpha of 0.05, a power of 0.80, and a 1:1 group allocation, the calculated minimum sample size required for significance is 349 infants for each arm, leading to a total of N=698 infants. Accounting for an estimated 5% dropout rate during follow-up, the adjusted minimum sample size becomes N=736 infants"

DATA ANALYSIS:

Data will be analysed according to an intention-to-treat model. Therefore, data from all infants enrolled into the study will be considered for the analysis. Death and transfer to another hospital before discontinuation of infusion therapy, are the only two reasons for exclusion. The primary outcome will be evaluated by Fisher's exact test. Secondary outcomes will be evaluated by Fisher's exact test or appropriate generalized linear models.

EXPECTED RESULTS AND IMPACT ON CLINICAL PRACTICE:

If the use of in-line filters resulted in a significant decrease in negative-culture inflammatory episodes and/or in any other complications, the use of in-line filters in all intravenous administration systems may be recommended in NICU.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to NICU with at least one central venous catheter

Exclusion Criteria:

* Patients with peripheral venous catheter, patients with inflammatory episode at the time of enrollment

Ages: 1 Hour to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 736 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Frequency of patients with at least one inflammatory episode sepsis-like. | From date of randomization until the date of hospital discharge or date of death, whichever came first, assessed up to 6 months
  Frequency of patients with at least one inflammatory episode sepsis-like, defined by alteration of the biomarkers of inflammation in a negative-culture contest.

SECONDARY OUTCOMES:
Frequency of patients with at least one episode of sepsis. | From date of randomization until the date of hospital discharge or date of death, whichever came first, assessed up to 6 months
  Frequency of patients with at least one inflammatory episode defined by alteration of the biomarkers of inflammation in a positive-culture contest.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Cresi, PhD MD, Study Director — University of Turin, Italy; Alessandra Coscia, PhD MD, Study Director — University of Turin, Italy; Elena Maggiora, MD, Principal Investigator — University of Turin, Italy; Cecilia Capetti, MD, Principal Investigator — University of Turin, Italy; Francesca De Matteis, RN, Principal Investigator — Città della salute e della Scienza di Torino; Martina Capitanio, MD, Principal Investigator — University of Turin, Italy; Fabio Mosca, Prof., Study Chair — University of Milan, Italy
Locations (1):
- Città della Salute e della Scienza, Torino, Italia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van den Hoogen A, Krediet TG, Uiterwaal CS, Bolenius JF, Gerards LJ, Fleer A. In-line filters in central venous catheters in a neonatal intensive care unit. J Perinat Med. 2006;34(1):71-4. doi: 10.1515/JPM.2006.009. PMID 16489888
- [Background] Sasse M, Dziuba F, Jack T, Koditz H, Kaussen T, Bertram H, Beerbaum P, Boehne M. In-line Filtration Decreases Systemic Inflammatory Response Syndrome, Renal and Hematologic Dysfunction in Pediatric Cardiac Intensive Care Patients. Pediatr Cardiol. 2015 Aug;36(6):1270-8. doi: 10.1007/s00246-015-1157-x. Epub 2015 Apr 7. PMID 25845941
- [Background] Virlouvet AL, Pansiot J, Toumazi A, Colella M, Capewell A, Guerriero E, Storme T, Rioualen S, Bourmaud A, Biran V, Baud O. In-line filtration in very preterm neonates: a randomized controlled trial. Sci Rep. 2020 Mar 19;10(1):5003. doi: 10.1038/s41598-020-61815-4. PMID 32193413
- [Background] Jack T, Boehne M, Brent BE, Hoy L, Koditz H, Wessel A, Sasse M. In-line filtration reduces severe complications and length of stay on pediatric intensive care unit: a prospective, randomized, controlled trial. Intensive Care Med. 2012 Jun;38(6):1008-16. doi: 10.1007/s00134-012-2539-7. Epub 2012 Apr 12. PMID 22527062
- [Background] Foster JP, Richards R, Showell MG, Jones LJ. Intravenous in-line filters for preventing morbidity and mortality in neonates. Cochrane Database Syst Rev. 2015 Aug 6;2015(8):CD005248. doi: 10.1002/14651858.CD005248.pub3. PMID 26244380
- [Background] Eschborn S, Weitkamp JH. Procalcitonin versus C-reactive protein: review of kinetics and performance for diagnosis of neonatal sepsis. J Perinatol. 2019 Jul;39(7):893-903. doi: 10.1038/s41372-019-0363-4. Epub 2019 Mar 29. PMID 30926891
- [Background] van Lingen RA, Baerts W, Marquering AC, Ruijs GJ. The use of in-line intravenous filters in sick newborn infants. Acta Paediatr. 2004 May;93(5):658-62. doi: 10.1111/j.1651-2227.2004.tb02993.x. PMID 15174791
- [Background] Worthington P, Gura KM, Kraft MD, Nishikawa R, Guenter P, Sacks GS; ASPEN PN Safety Committee. Update on the Use of Filters for Parenteral Nutrition: An ASPEN Position Paper. Nutr Clin Pract. 2021 Feb;36(1):29-39. doi: 10.1002/ncp.10587. Epub 2020 Oct 22. PMID 33091206
- [Derived] Cresi F, Maggiora E, Capetti C, Capitanio M, Ferroglio M, Spada E, De Matteis F, Cosimi S, Mosca F, Coscia A; INCAS Trial Research Group. Effect of in-line filtration in newborns: study protocol of the Intravenous Neonatal Central Access Safety (INCAS) randomized controlled trial. Trials. 2024 Jul 6;25(1):459. doi: 10.1186/s13063-024-08264-w. PMID 38971756